CLINICAL TRIAL: NCT02729636
Title: Multi-pad Functional Electrical Stimulation for Droop Foot Treatment
Brief Title: Multi-pad FES System for Drop Foot Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Konstantinovic Ljubica, professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LK-4
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Foot Drop
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FES:a (Experimental): The group will be treated with multipad electrical stimulation device.
  Interventions: Device: multi-pad functional electrical stimulation (FES)
- control (Active Comparator): The group will be treated with conventional treatment.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: multi-pad functional electrical stimulation (FES) — Treatment includes two automated phases: optimization of stimulation parameters and application during the walk.
  Optimization of stimulation parameters: The stimulator generates short bursts of electrical impulses and sends them to each of the 16 pads of the multi-pad electrode. Each pad is the same size. Pads are sorted in two rows by 8 pads. Common anode is placed under the knee. Based on FES-induced foot movements, automated algorithm suggests parameters which are evaluated by medical doctor/therapist.
  Assisted walking: During assisted walking, pattern for plantar flexion is activated in push off phase and pattern for dorsiflexion in swing phase of the gait.
  Arms: FES:a
Other: Conventional therapy — 2. All study subjects received the conventional stroke rehabilitation program of physiotherapy based on the neurodevelopmental facilitation approach and occupational therapy focused on activities of daily living during the treatment for 60 min a day, 5 days a week, for 4-weeks. Conventional therapy was given by trained therapists and consisted of the following strategies: strategies to joint mobilization and range of motion exercises; exercises to improve strength; strategies to manage spasticity; exercises for increase range of motion, compensatory strategy; strategies to improve balance, and mobility.
  Arms: control

SUMMARY:
Functional electrical stimulation (FES) is multi-pad system that allows fast optimization of stimulation patterns for achieving strong dorsiflexion/plantar flexion and automatic real-time control of ankle joint during FES assisted walking. The main aim of the present study is to compare the effects of functional electrical stimulation gait training after stroke and overground conventional physical therapy. With the assumption that the advanced method of functional electrical stimulation will improve gait parameters and functionality in patients with foot drop before and after FES treatment the objectives of this study are to examine the effects of functional electrical stimulation using FES:a method on indicators of walk and function in patients with foot drop before and after FES treatment.

ELIGIBILITY:
Inclusion Criteria:

* hemiplegia caused by stroke
* inadequate ankle dorsiflexion
* passive ankle range of motion to neutral position
* adequate cognitive and communication function to give informed consent
* sufficient motor ability and endurance to ambulate at least 6 minutes of walking independently with or without an assistive device
* calf muscle spasticity not higher than grade 3 according to the Modified Ashworth Scale

Exclusion Criteria:

* lower motor neuron injury with inadequate response to stimulation
* skin rupture in the area of the electrodes
* history of falls greater than once a week
* multiple or infratentorial cerebrovascular lesions
* severe cardiovascular disease, severe auditory and visual impairments
* inadequate response to stimulation (range of motion elicit by maximal pleasant stimulation lower than active range in first 5 days of the therapy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
gait speed by 10m walking test | 4 weeks

SECONDARY OUTCOMES:
motor arm impairment by Fugl Mayer assessment | 4 weeks
Activities of daily living by Barthel index | 4 weeks
postural stability by Berg Balance scale | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for rehabilitation dr Miroslav Zotovic Faculty of Medicine University of Belgrade, Belgrade, Serbia

REFERENCES:
- [Derived] Malesevic J, Dedijer Dujovic S, Savic AM, Konstantinovic L, Vidakovic A, Bijelic G, Malesevic N, Keller T. A decision support system for electrode shaping in multi-pad FES foot drop correction. J Neuroeng Rehabil. 2017 Jul 3;14(1):66. doi: 10.1186/s12984-017-0275-5. PMID 28673311